CLINICAL TRIAL: NCT02426333
Title: Optimizing Abiraterone (Zytiga®) Therapy by Exploring the Relation Between an Early Biomarker - Drug Exposure - as a Predictor for Drug Response in Patients With mCRPC
Brief Title: Optimizing Abiraterone Therapy
Acronym: OPTIMUM
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: UMCN AKF-14.07
Record Dates: First submitted 2015-03-27; First posted 2015-04-24 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for abiraterone concentrations and also blood samples to assess biomarkers (some contain DNA)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abiraterone Acetate: abiraterone treatment, 1000mg, tablets, once daily, treatment is not adapted for the study
  Interventions: Other: Abiraterone Acetate

INTERVENTIONS:
Other: Abiraterone Acetate — Exclusively determine pharmacokinetics and pharmacodynamics of abiraterone for the indication according to the drug label (CRPC)

SUMMARY:
The purpose of this study is to explore whether early abiraterone exposure is related to treatment response in patients with metastatic castration resistant prostate cancer. Furthermore to explore the relation between biomarkers and treatment response and drug exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic castration resistant prostate cancer who are asymptomatic or mildly symptomatic after failure of androgen deprivation therapy in whom chemotherapy is not yet clinically indicated
* Age ≥18 years
* Feasible to collect blood samples from
* Life expectancy of > 6 months
* Measurable disease
* Able and willing to give written informed consent prior to screening and enrollment

Exclusion Criteria:

* other anticancer therapies
* potent CYP3A4 inducers
* herbal medicine that could interfere with abiraterone exposure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with metastatic castration resistant prostate cancer who are asymptomatic or mildly symptomatic after failure of androgen deprivation therapy in whom chemotherapy is not yet clinically indicated
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
abiraterone AUC | 6 months

SECONDARY OUTCOMES:
biomarkers: relation between biomarkers and treatment response | 6 months
  relation between biomarkers and treatment response
biomarker reduction | 6 months
  To explore the if reduction in biomarkers is related to treatment response after three and six months

CONTACTS AND LOCATIONS:
Overall Officials: Nielka van Erp, PharmD, PhD, Principal Investigator — Radboud University Medical Center; Jack Schalken, PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud UMC, Nijmegen

IPD SHARING:
Plan to Share IPD: No